CLINICAL TRIAL: NCT06519994
Title: Feasibility of Intravaginal Artesunate as Adjuvant HPV & Cervical Precancer Treatment Among Women Living With HIV in Kenya
Brief Title: Feasibility of Intravaginal Artesunate as Adjuvant HPV & Cervical Precancer Treatment in Kenya
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Kenya Medical Research Institute (Other); Maseno University School of Medicine, Kenya (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCCC2330; R34CA284983 (NIH)
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Human Immunodeficiency Virus; Human Papillomavirus; Cervical Precancer
Keywords: intravaginal; self-administer; artesunate; intravaginal artesunate; vaginal pessaries
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artesunate vaginal inserts (Experimental): Participants will self-administer the study drug nightly for 5 days, take a week off, and repeat 2 times (study drug application on weeks 1, 3, 5).
  Interventions: Drug: Artesunate vaginal inserts
- Placebo vaginal inserts (Placebo Comparator): Participants will self-administer the study placebo nightly for 5 days, take a week off, and repeat 2 times (study drug application on weeks 1, 3, 5).
  Interventions: Drug: Placebo vaginal inserts

INTERVENTIONS:
Drug: Artesunate vaginal inserts — Subjects will self-administer 200 mg of Artesunate vaginal insert daily for 5 days, on weeks 1, 3, 5.
  Arms: Artesunate vaginal inserts
Drug: Placebo vaginal inserts — Subjects will self-administer a placebo vaginal insert daily for 5 days, on weeks 1, 3, 5.
  Arms: Placebo vaginal inserts

SUMMARY:
The objective of this randomized, placebo-controlled trial is to evaluate whether intravaginal artesunate pessaries (vaginal inserts) can be used as adjuvant therapy following thermal ablation to improve Human papillomavirus (HPV) treatment outcomes in Women Living with Human Immunodeficiency Virus (WLWH).

The study will evaluate whether women who use artesunate will have higher HPV clearance at 6 months, compared to those who used a placebo. The study will also assess the safety, adherence, and acceptability of this treatment. 120 participants will be enrolled in the study. Participants will self-administer the study drug nightly for 5 days, take a week off, and repeat twice (use study drug on weeks 1, 3,5) and will return to the clinic on weeks 2, 4, 6, 12, and week 24 for follow-up.

DETAILED DESCRIPTION:
WLWH face up to six times increased risk of cervical cancer, as a result, cervical cancer is a leading cause of death in this population. Cervical cancer is caused by persistent infection with the human papillomavirus (HPV), resulting in precancerous changes that if not adequately treated, progress to cancer. Thermal ablation is a commonly used treatment for cervical precancer in Kenya and other low- and middle-income countries (LMICs). Current treatments for HPV or cervical precancer, including thermal ablation, are associated with high rates of treatment failure in WLWH. In a recent study from Zambia, only 44% of WLWH had cleared HPV at six months following thermal ablation treatment. Other studies have demonstrated up to 30% recurrence rate of high-grade cervical precancer at 12 to 24 months after treatment. Persistent infection with HPV following precancer treatment is a key risk factor for treatment disease recurrence.

ELIGIBILITY:
Inclusion Criteria

* Age 25 years or older
* Known HIV seropositive status
* On antiretroviral therapy for > 90 days prior to enrollment
* Weight ≥50 Kg at study entry*
* Positive HPV screening test and within 4-8 weeks of thermal ablation
* Ability to provide informed consent
* Planning to stay within the study locale during the duration of the study (24 weeks)
* Agreement to use contraception (barriers or hormonal) if of childbearing age through week 6 of the study

Exclusion Criteria

* Current pregnancy or breastfeeding status
* Current or past history of invasive cervical cancer
* History of total hysterectomy
* Currently receiving systemic chemotherapy or radiation therapy for another cancer
* Current use of systemic immunosuppressants or steroids (>10 mg of prednisone or equivalent)
* Current use of efavirenz antiretroviral therapy, phenytoin, carbamazepine, and rifampin
* Have medical comorbidity that, in the opinion of the investigator, would interfere with study participation
* Prior chemotherapy within 30 days prior to day 1 of study treatment
* Male at birth

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned biological female gender at birth.
Enrollment: 120 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Clearance of type-specific HPV genotype(s) | 24 weeks
  The number and proportion of women in each study arm who demonstrate clearance of the specific HPV genotype, or genotypes (if multiple) between baseline and six months will be reported.

SECONDARY OUTCOMES:
Adherence | Week 6
  Adherence will be evaluated based on the number and proportion of women confirmed self-administration of at least 80% (12 of 15) vaginal inserts.
Acceptability measured by acceptability questionnaire | Week 6
  Acceptability will be evaluated based on a close-ended structured acceptability questionnaire. The responses will be on a Likert score, between 1-5, and higher scores represent better accepted.

OTHER OUTCOMES:
Uptake | Baseline
  Number of screen-eligible participants who agree to enroll in the study.
Accrual rate | 24 weeks
  Number of participants that enrolled in the trial divided by time from the first enrollment to the last enrollment in months.
Retention rate | 24 weeks
  Retention rate: Number of women in each study arm retained in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Chemtai Mungo, MD, MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lumumba Sub-County Hospital KEMRI- Research Care Training Program (RCTP) Building, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sadana A, Omoto J, Sorgi K, Rahangdale L, Smith JS, Plesa M, Mungo C. Feasibility of Intravaginal Artesunate as an Adjuvant HPV & Cervical Precancer Treatment Among Women Living With HIV in Kenya: Study Protocol for a Phase II Clinical Trial. Cancer Control. 2025 Jan-Dec;32:10732748251374418. doi: 10.1177/10732748251374418. Epub 2025 Sep 4. PMID 40907021
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials